CLINICAL TRIAL: NCT05221905
Title: Effects of Inorganic Nitrate and Intensity of Exercise on Cardiovascular Health in Post-Menopausal Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Arthur L Weltman, Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HSR210326
Record Dates: First submitted 2021-10-14; First posted 2022-02-03 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Vascular Dilation; Arterial Stiffness
Keywords: Flow-mediated dilation; Pulse wave velocity; Exercise intensity; Vascular function

STUDY DESIGN:
Intervention Model Description: Subject are stratified randomized to consume either beetroot juice with, or without, inorganic nitrate and will consume this same supplement throughout all testing
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study, where neither the investigators nor the subjects will know whether the participants are receiving the active supplement or placebo supplement until study conclusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Acute High-Intensity Exercise (Active Comparator): Subjects will exercise at an intensity of 75% of the difference between the lactate threshold and VO2peak until 200 kcal are expended. Pre- and post-testing measures of vascular health will be completed at baseline (0 min) and again 60, 90, 120, 150, 180 min post-baseline testing, with exercise taking place during time points 0-60 min.
  Interventions: Drug: BEET IT - Concentrate Beet root juice; Drug: BEET IT - Concentrate Beet root juice (nitrate depleted)
- Acute Moderate-Intensity Exercise (Active Comparator): Subjects will exercise at an intensity at the lactate threshold until 200 kcal are expended. Pre- and post-testing measures of vascular health will be completed at baseline (0 min) and again 60, 90, 120, 150, 180 min post-baseline testing, with exercise taking place during time points 0-60 min.
  Interventions: Drug: BEET IT - Concentrate Beet root juice; Drug: BEET IT - Concentrate Beet root juice (nitrate depleted)
- Non-Exercise Control (Placebo Comparator): Measures of vascular health will be completed at baseline (0 min) and again 60, 90, 120, 150, 180 min post-baseline testing, without exercise taking place during time points 0-60 min.
  Interventions: Drug: BEET IT - Concentrate Beet root juice; Drug: BEET IT - Concentrate Beet root juice (nitrate depleted)

INTERVENTIONS:
Drug: BEET IT - Concentrate Beet root juice — Beet It Sport (James White Drinks, Ltd.) each containing 400mg of inorganic nitrate (~6.5 mmol) will be consumed twice daily (totalling ~13 mmol of inorganic nitrate per day) for at least 2 days prior to testing visits, as well as 2 hours prior to testing visits.
  Other Names: Dietary Nitrate supplementation (nitrate rich)
Drug: BEET IT - Concentrate Beet root juice (nitrate depleted) — Beet It Sport (James White Drinks, Ltd.) each containing 0mg of inorganic nitrate (~0 mmol) will be consumed twice daily (totalling ~0 mmol of inorganic nitrate per day) for at least 2 days prior to testing visits, as well as 2 hours prior to testing visits. It is provided by the same company that produces the concentrated beet root juice shots (James White Drinks) but the placebo version is nitrate-depleted.
  Other Names: Dietary Nitrate supplementation (nitrate depleted)

SUMMARY:
Post-menopausal females experience elevated cardiovascular disease risk (CVD), compared to premenopausal females and age-matched males. Current exercise guidelines appear inadequate to ameliorate this increased risk and higher intensity exercise may be necessary. Oral inorganic nitrate supplementation enhances both exercise performance and CVD risk profile in several clinical conditions. However, the effects of this intervention in post-menopausal females is unexplored.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether acute inorganic nitrate supplementation and exercising at different exercise intensities (high vs moderate) improve vascular health in post-menopausal females.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal female, defined as having not had a menstrual cycle for at least 1 year
* Greater than age 45 but less than age 75
* Sedentary (does not exercise regularly)
* No major changes in medication in the last 3 months

Exclusion Criteria:

* Smokers within last 5 years
* Weight unstable (loss/gain of more than 3kg in the past 3 months)
* Any medical condition that prevents the subject from exercising safely
* Hormone replacement therapy (current or within last 3 months)
* Currently or recently on vasoactive medications (i.e., calcium channel blockers, statins, ACE or renin inhibitors, ARBs, nitrates, alpha- or beta-blockers, diuretics, proton pump inhibitors, etc.)
* Hysterectomy or oophorectomy

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All subjects are post-menopausal females.
Enrollment: 24 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Baseline Flow-Mediated Dilation | Baseline (minute 0).
  Participants will be placed in a supine position with their left forearm slightly extended and supinated with legs straight. The brachial artery will be imaged using a high-resolution doppler ultrasound utilizing a 7.5MHz linear array transducer at rest, during 5 minutes of forearm occlusion via cuff inflation, and continuously for 2 minutes post-occlusion; an EKG trigger will be used to capture images during end-diastole of the cardiac cycle. Images will be analyzed offline using specialized software (Medical Imaging Applications, Inc.) to calculate the change in brachial artery diameter.
Post-Exercise/Control Flow-Mediated Dilation (60 minutes) | 60 minutes post-baseline.
  Participants will be placed in a supine position with their left forearm slightly extended and supinated with legs straight. The brachial artery will be imaged using a high-resolution doppler ultrasound utilizing a 7.5MHz linear array transducer at rest, during 5 minutes of forearm occlusion via cuff inflation, and continuously for 2 minutes post-occlusion; an EKG trigger will be used to capture images during end-diastole of the cardiac cycle. Images will be analyzed offline using specialized software (Medical Imaging Applications, Inc.) to calculate the change in brachial artery diameter.
Post-Exercise/Control Flow-Mediated Dilation (90 minutes) | 90 minutes post-baseline.
  Participants will be placed in a supine position with their left forearm slightly extended and supinated with legs straight. The brachial artery will be imaged using a high-resolution doppler ultrasound utilizing a 7.5MHz linear array transducer at rest, during 5 minutes of forearm occlusion via cuff inflation, and continuously for 2 minutes post-occlusion; an EKG trigger will be used to capture images during end-diastole of the cardiac cycle. Images will be analyzed offline using specialized software (Medical Imaging Applications, Inc.) to calculate the change in brachial artery diameter.
Post-Exercise/Control Flow-Mediated Dilation (120 minutes) | 120 minutes post-baseline.
  Participants will be placed in a supine position with their left forearm slightly extended and supinated with legs straight. The brachial artery will be imaged using a high-resolution doppler ultrasound utilizing a 7.5MHz linear array transducer at rest, during 5 minutes of forearm occlusion via cuff inflation, and continuously for 2 minutes post-occlusion; an EKG trigger will be used to capture images during end-diastole of the cardiac cycle. Images will be analyzed offline using specialized software (Medical Imaging Applications, Inc.) to calculate the change in brachial artery diameter.
Post-Exercise/Control Flow-Mediated Dilation (150 min) | 150 minutes post-baseline.
  Participants will be placed in a supine position with their left forearm slightly extended and supinated with legs straight. The brachial artery will be imaged using a high-resolution doppler ultrasound utilizing a 7.5MHz linear array transducer at rest, during 5 minutes of forearm occlusion via cuff inflation, and continuously for 2 minutes post-occlusion; an EKG trigger will be used to capture images during end-diastole of the cardiac cycle. Images will be analyzed offline using specialized software (Medical Imaging Applications, Inc.) to calculate the change in brachial artery diameter.
Post-Exercise/Control Flow-Mediated Dilation (180 min) | 180 minutes post-baseline.
  Participants will be placed in a supine position with their left forearm slightly extended and supinated with legs straight. The brachial artery will be imaged using a high-resolution doppler ultrasound utilizing a 7.5MHz linear array transducer at rest, during 5 minutes of forearm occlusion via cuff inflation, and continuously for 2 minutes post-occlusion; an EKG trigger will be used to capture images during end-diastole of the cardiac cycle. Images will be analyzed offline using specialized software (Medical Imaging Applications, Inc.) to calculate the change in brachial artery diameter.

SECONDARY OUTCOMES:
Baseline Pulse Wave Velocity | Baseline (minute 0).
  Supine measures of carotid to femoral pulse wave velocity will be measured using a SphygmoCor Xcel device.
Post-Exercise/Control Pulse Wave Velocity (60 min) | 60 minutes post-baseline.
  Supine measures of carotid to femoral pulse wave velocity will be measured using a SphygmoCor Xcel device.
Post-Exercise/Control Pulse Wave Velocity (90 min) | 90 minutes post-baseline.
  Supine measures of carotid to femoral pulse wave velocity will be measured using a SphygmoCor Xcel device.
Post-Exercise/Control Pulse Wave Velocity (120 min) | 120 minutes post-baseline.
  Supine measures of carotid to femoral pulse wave velocity will be measured using a SphygmoCor Xcel device.
Post-Exercise/Control Pulse Wave Velocity (150 min) | 150 minutes post-baseline.
  Supine measures of carotid to femoral pulse wave velocity will be measured using a SphygmoCor Xcel device.
Post-Exercise/Control Pulse Wave Velocity (180 min) | 180 minutes post-baseline.
  Supine measures of carotid to femoral pulse wave velocity will be measured using a SphygmoCor Xcel device.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Weltman, PhD, Principal Investigator — Professor of Kinesiology
Locations (1):
- Student Health and Wellness Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Microsoft excel sheets, Graphpad Prism files, Informed Consent, and Study Protocol forms will be available upon reasonable request. All identifiable data de-identified on 24 participants will be available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified data will be shared upon reasonable request for 3 years after study completion
Access Criteria: Email Austin Hogwood at ach2jb@virginia.edu for any requests.